CLINICAL TRIAL: NCT03284138
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of First Rank Symptoms on Schizophrenia: Controlled, Randomised, Double Blind Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of First Rank Symptoms (FRS) on Schizophrenia
Acronym: Schirang
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P150906
Record Dates: First submitted 2017-09-06; First posted 2017-09-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia Patients With First Rank Symptoms
Keywords: Schizophrenia; rTMS; first rank symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS treatment (Active Comparator): patient will be treated with 10 sessions in 5 days with low frequency (1Hz) of Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: rTMS treatment
- Placebo treatment (Sham Comparator): patient will be treated with 10 sessions in 5 days with low frequency (1Hz) of Sham-controlled
  Interventions: Device: placebo treatment

INTERVENTIONS:
Device: rTMS treatment — patient will be treated with 10 sessions in 5 days with low frequency (1Hz) of Repetitive Transcranial Magnetic Stimulation (rTMS)
  Other Names: intervention
  Arms: rTMS treatment
Device: placebo treatment — patient will be treated with 10 sessions in 5 days with low frequency (1Hz) of Sham-controlled
  Other Names: placebo
  Arms: Placebo treatment

SUMMARY:
First rank symptoms are core symptoms of schizophrenia. the investigators want to offer an integrative approach to better understanding of the mechanisms involved in the first rank symptoms and therefore, in schizophrenia, as well as the neuronal modulation mechanisms obtained by rTMS. It will be to pass a functional magnetic resonance imaging (fMRI) at rest for healthy volunteers, and for patients before and after rTMS modulation, to view brain structures activated in the resting state network, and in order to study

1. the difference of the resting-state network between healthy volunteers and people with schizophrenia,
2. if the response to rTMS boost can be predicted by resting-state network of patients before treatment and
3. if rTMS changes activations in the brain of patients. This will ultimately provide rTMS as a treatment of first rank symptoms.

DETAILED DESCRIPTION:
Schizophrenia is a common psychiatric disorder that affects approximately 1% of the general population. This disease can be described in three dimensions: disorganization, delusions and negative signs. The "first rank symptoms" (FRS) were first described by Kurt Schneider. These are core symptoms of schizophrenia that were combined to make pathognomonic signs of the disease and remain at the center of many classifications of the disease. These symptoms are voices or thoughts expressed aloud, voices who argue them, voices that comment on behavior or thoughts, delusional perceptions, experiences of body influences, thoughts influences, impulses from external influences, the will controlled by external forces, thoughts stolen by external forces or others, thoughts interferences by other thoughts, publication thoughts. These symptoms reveal difficulty in distinguishing self and other in action, thought or physical individual. Thus, the FRS are a gateway to agency disorder, disorder of the sense of body ownership and familiarity disorder.

Agency is the ability to distinguish ones own actions from those of others. The sense of body ownership is difficult to distinguish from the sense of agency. It is the knowledge that the arm (for example) which make this action is mine. A disorder of sense of body ownership may lead to the illusion of a phantom limb and it is very interesting to separate both mechanisms of body ownership and agency as wall as the networks involved in agency of those involved in the sense of body ownership. Familiarity is the feeling associated with the sight of someone close. Thus, in familiarity disorder, patient recognizes the facial features of relatives, but feels no sense of familiarity and attributes this to the replacement of the close by an impostor. Familiarity disorders can be understood through the 2-ways model of faces of processing in which the ventral pathway would be affected in the familiarity disorder. The ventral pathway involves a network which extends from the visual cortex to the superior temporal sulcus, the inferior parietal lobe and the cingulate gyrus to join the dorsal pathway in the hypothalamus.

In addition, agency studies imply the superior temporal sulcus and the inferior parietal lobule as regions involved in distinguishing self / others. Nowadays, remains a difficulty to clearly identify the different functions of the regions involved in agency.

Few neuroimaging studies can identify key areas of the sense of body ownership; in fact, protocols are difficult to adapt for use in a scanner. However, there are few studies that highlight, as was expected, extrastriatal body area as well as areas that may be involved in agency. Experiments have difficulty differentiating, as the investigators said, the sense of body ownership from agency, but the investigators have a validated tool, the rubber hand illusion, to differentiate sense of body ownership and agency. This tool has already been validated in healthy subjects , and was the subject of a study in our unit on patients with schizophrenia about to be published. In addition, several studies have shown that the performance at the rubber hand illusion task were modified by repeated Transcranial Magnetic Stimulation (rTMS) applied to the extrastriatal body area (EBA) or to the inferior parietal lobule (IPL) or to the temporo-parietal junction (TPJ).

Transcranial magnetic stimulation or TMS modulate cortical excitability without serious side effects when used at frequencies and intensities recommended in the literature. Low frequency rTMS is a recognized for treatment-resistant auditory hallucinations in schizophrenia. This is therefore an interesting therapeutic innovation that will benefit to residual symptoms, in adjunction to a well conducted medical treatment in schizophrenia.

To our knowledge, no study has been performed using rTMS as a treatment for FRS in schizophrenia. The investigators propose to evaluate the impact of treatment with low-frequency rTMS applied to the superior temporal sulcus in its posterior part (pSTS) on disorders of agency and familiarity. Indeed, it is well established that low-frequency rTMS (1 Hz) of the left TPJ was used to reduce auditory hallucinations in schizophrenia. On the same model, the investigators want to offer an innovative and integrative treatment of core symptoms of schizophrenia with the specificity of not focusing on a single symptom. The choice of pSTS allows also operating on the sense of body ownership inasmuch the TPJ is adjacent to the pSTS.

In addition, in order to have a more comprehensive study incorporating different aspects of the pathophysiology of schizophrenia, the investigators want to add a functional magnetic resonance imaging (fMRI) of resting-state. This would be to pass a fMRI for healthy volunteers. For people with schizophrenia, they will pass a fMRI before and after treatment for visualizing brain structures activated in the resting-state network, in order to study

1. the difference in resting-state circuitry between healthy volunteers and schizophrenia patients
2. whether the response to treatment with rTMS could be predicted by resting-state network of patients before treatment and
3. whether treatment with rTMS could modulate brain activations of patients.

Indeed, the resting-state network is the brain activity that occurs when a subject leaves his mind at rest without any particular task. Self-awareness is involved in this resting-state network. This network involves bilateral structures with the main nodes in medial prefrontal cortex, posterior cingulate cortex, precuneus and angular gyrus. People with schizophrenia exhibit connectivity anomalies in the resting-state network that are temporal connection anomalies. In acoustico-verbal hallucinations, people with schizophrenia have a resting-state network particularly active in the auditory cortex. Authors have proposed that this hyperactivity of the auditory cortex in the resting-state network would make patients more vulnerable to attribute external stimuli to them.

Similarly, it can be postulated that patients with FRS would have a hyperactivity of the resting-state network especially in the pSTS and the TPJ, which would lead to a difficulty in distinguishing oneself and others and thus, to FRS. Thus, the investigators hypothesize that patients with abnormal functional connectivity in the resting-state network (mainly in the pSTS and TPJ, which the investigators will then be boost in rTMS) will have a better response to treatment and that, after rTMS treatment, a change will be visible on neuronal activation of resting-state network in fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from schizophrenia (according to DSM IV-TR)
* Presenting FRS at least once a day despite well-conducted antipsychotic treatment, objectified by FRS subscore of the SAPS (items 2, 3 and items 15-19) with at least two FRS listed > 1 of the corresponding item of the SAPS
* Being informed of the objectives and constraints of the study and signing the consent form or signing by the guardian
* Patient having had a preliminary clinical examination

Exclusion Criteria:

* Left-lateralized
* Previously treated with rTMS in the previous 6 month,
* Contraindications of the rTMS practice: unstabilized epilepsy, presence of foreign eye metallic material, pacemaker, neurostimulator, cochlear implants and in general all medical equipment installed immovably, metal heart valve, vascular clips formerly located on cranial aneurysm
* Pregnancy or breastfeeding women
* hospitalization under constraint
* Subject already involved in another interventional clinical research evaluating schizophrenia treatment
* patient with severe drug use disorder (excluding coffee and tobacco) according to the DSM-5 criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of first rank symptoms | 5 days after inclusion
  Number of first rank symptoms measured by items 2,3 and 15 to 19 of "first rank" subscore from SAPS

SECONDARY OUTCOMES:
Evaluation of both agency and sense of body ownership disorders with Rubber Hand Illusion test (RHI) | 5 days, 1 month and 3 months after inclusion
  RHI Test is composite evaluation . A wooden hand will be placed in front of the subject while his proper hand rests, hidden from his vision. When applying identical and synchronous active movement to both the wooden and the subject hidden hand, subject feels rapidly as moving directly to the rubber hand level, and develops a sense of ownership to this artificial hand.
  1. The intensity of the illusion is measured subjectively by answering a questionnaire (over sense of one's own body and agency).
  2. The intensity of the illusion is measured objectively by measuring proprioceptive bias in millimeters after each stimulation by asking the subject to place his own hand after illusion induction.
Evaluation of familiarity disorder | 5 days, 1 and 3 month after inclusion
  Face morphing tasks have been used for a decade to identify facial recognition defects and allow calculating a recognition threshold (percentage of the faces morphed required for recognition). This threshold may be compared over time. Faces are morphed between the subject's face with same sex pictures either familiar (2 persons close to the patient) or unfamiliar (two faces from a database34). The subjects indicate when they recognize their relative or when a stranger emerges during computer presentation of morphed images, to a varying extent from 0 to 100% (by 10% step). A threshold of recognition per conditions (self, familiar, unknown) will be extract for each subject as a percentage
Evaluation of the severity of symptoms | 5 days, 1 and 3 month after inclusion
  use of the Positive And Negative Symptoms Scale PANSS, an hetero evaluation of schizophrenia symptoms
Evaluation of the functioning | 5 days, 1 and 3 month after inclusion
  By using the Global Assessment of Functioning (GAF)
Evaluation of quality of life | 5 days, 1 and 3 month after inclusion
  By using the Shortened Quality of Life Questionnaire (S-QoL 18)
Evaluation of the side effects | 5 days after inclusion
  By using the Side effects surveillance (UKU)

CONTACTS AND LOCATIONS:
Overall Officials: Aurely Ameller, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Louis Mourier, Colombes, France

IPD SHARING:
Plan to Share IPD: Undecided